CLINICAL TRIAL: NCT00221598
Title: Effect of Dialysate Temperature on Haemodynamic Stability and Haemodialysis Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005/148
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Acute Renal Failure; Chronic Renal Failure
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemodialysis (Experimental)
  Interventions: Procedure: Haemodialysis with different dialysate temperatures

INTERVENTIONS:
Procedure: Haemodialysis with different dialysate temperatures — Haemodialysis with different dialysate temperatures is used.

SUMMARY:
Comparison between dialysate temperatures on haemodynamic stability and haemodialysis efficiency.

DETAILED DESCRIPTION:
Comparison of 4 different dialysate temperatures for haemodialysis of patients with chronic renal failure.

Comparison of 3 different dialysate temperatures for haemodialysis of patients with acute renal failure.

Investigation of the efficiency of haemodialysis of patients with acute renal failure

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure
* Acute renal failure
* Aged between 21-90 years

Exclusion Criteria:

-

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2010-12-14 (Actual)

PRIMARY OUTCOMES:
Haemodynamic stability and tolerance | t0

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Dhondt, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be